CLINICAL TRIAL: NCT03128723
Title: A Single Center Clinical Study to Evaluate the Tolerance of an Acne Treatment in Sensitive Skin Subjects With Mild to Moderate Acne Vulgaris
Brief Title: A Study to Evaluate the Tolerance of an Acne Treatment in Sensitive Skin Subjects With Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-170125113728-SACT
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Acne Mask (Experimental): The light therapy acne mask is applied to the face once in the evening for a duration of 10 minutes. The cleanser is used twice daily, once in the morning and once in the evening.
  Interventions: Device: Acne Mask

INTERVENTIONS:
Device: Acne Mask — The light therapy acne mask contains a combination of red and blue light-emitting diodes. The device is applied once daily, in the evening for a duration of 10 minutes.
  Other Names: Light Therapy Acne Mask

SUMMARY:
The study will look to evaluate the tolerance of a light therapy-based acne mask device in participants who report having sensitive skin. All participants will receive a cleanser, a light therapy mask, and an extra activator for the light therapy mask.

DETAILED DESCRIPTION:
Acne and sensitive skin can be closely connected due to the reported involvement of an impaired skin barrier in both conditions, which can be further aggravated by potentially irritating topical treatments.

A patient's sensitive skin may be caused by the skincare products that they are using, the amount that they are applying (over-usage), or the concomitant effect of the different products being used, as well as by underlying medical conditions. While sensitive skin can be self-perceived and sometimes clinically apparent, as there is no agreed upon medical definition of 'sensitive skin', it is a 'diagnosis' primarily made by the patient's perception. The high incidence of this problem and potential for further irritation due to current topical treatments has left many patients in need of a sensitive skin solution for their acne.

Current at-home topical treatments for mild to moderate acne include Over-the-Counter (OTC) options, primarily with either benzoyl peroxide, or salicylic acid, as well as prescription options including retinoid-based products, however the cutaneous irritation potential of topical acne active ingredients has been reported in the literature, which is not desirable in particular for patients with sensitive skin.

Research has shown the benefits of red and blue light therapy in the treatment of mild to moderate acne, with blue light reported to target acne-causing bacteria and red light demonstrating anti-inflammatory activity. Previous studies with these types of modalities have shown high tolerance and efficacy. This study will look to evaluate the tolerance of a light therapy-based medical device in patients with self-reported sensitive skin.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Has mild to moderate facial acne
* Has sensitive skin per sensitive skin questionnaires
* Has score of "0" or "1" in all tolerance parameters (erythema, dryness/scaling, edema, burning/stinging, itching, and tightness/dryness feeling)
* Able to read, write, speak, and understand English
* Must agree to practice a medically acceptable form of birth control

Exclusion Criteria:

* Has known light or photo-sensitivity disorder
* Has very sensitive skin or known allergies to skincare products or the cleanser ingredients
* Has severe acne or pre-existing facial skin conditions other than mild to moderate acne
* Females that are pregnant, nursing, or planning to become pregnant
* Males with a female partner who is pregnant or planning to become pregnant
* Has been using a product or medication that the investigator determines will increase health risk to the subject or confuse the study results
* Is participating or has participated in another study with the past 30 days
* Has history of immunosuppression/immune deficiency disorders
* Has planned surgeries or invasive medical procedures scheduled during the study
* Is related to the Sponsor, Investigator, or Study Site

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Gold, M.D., Principal Investigator — Tennessee Clinical Research Center
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muizzuddin N, Marenus KD, Maes DH. Factors defining sensitive skin and its treatment. Am J Contact Dermat. 1998 Sep;9(3):170-5. PMID 9744910
- [Background] Willis CM, Shaw S, De Lacharriere O, Baverel M, Reiche L, Jourdain R, Bastien P, Wilkinson JD. Sensitive skin: an epidemiological study. Br J Dermatol. 2001 Aug;145(2):258-63. doi: 10.1046/j.1365-2133.2001.04343.x. PMID 11531788
- [Background] Sagransky M, Yentzer BA, Feldman SR. Benzoyl peroxide: a review of its current use in the treatment of acne vulgaris. Expert Opin Pharmacother. 2009 Oct;10(15):2555-62. doi: 10.1517/14656560903277228. PMID 19761357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 04, 2017, to May 10, 2017.
  Location: Clinical site.
Period: Overall Study
Arm/Group | Acne Mask
Started | 45
Completed | 43
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 30
  More than one race | 1
  Unknown or Not Reported | 1
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick skin type range I to VI:
  I: White; very fair; red or blonde hair; blue eyes; freckles; Always burns easily; never tans II: White; fair; red or blonde hair; blue hazel, or green eyes; Always burns easily; tans minimally III: Cream white; fair with any eye or hair color; very common; Burns moderately; tans gradually IV: Brown; typical Mediterranean white skin; Burns minimally; always tans well V: Dark brown; mid-eastern skin types, black hair, olive skin; Rarely burns; tans profusely VI: Black; black hair, black eyes, black skin; Never burns; deeply pigmented
  Participants
    I | 0
    II | 15
    III | 11
    IV | 6
    V | 4
    VI | 9
Investigator's global acne assessment [Count of Participants; unit: Participants] — Investigator's global acne assessment score 0-4
  Participants
    0 (clear) | 0
    1 (Almost clear) | 0
    2 (mild) | 28
    3 (moderate) | 17
    4 (severe) | 0
Do you consider your facial skin to be sensitive? [Count of Participants; unit: Participants]
  None of the time | 0
  Some of the time | 0
  Most of the time | 26
  All of the time | 19
In the past, have you ever experienced skin irritation when using topical acne treatments? [Count of Participants; unit: Participants]
  Yes | 38
  No | 7
In the past, have you ever stopped using a topical acne treatment due to skin irritation [Count of Participants; unit: Participants]
  Yes | 25
  No | 20
Have you ever been told by a skin care professional that you have sensitive skin on your face? [Count of Participants; unit: Participants]
  Yes | 15
  No | 30
When purchasing skincare products, do you look for products labeled "for sensitive skin" or similar? [Count of Participants; unit: Participants]
  Yes | 42
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Tolerance Scores: Erythema
Description: Cutaneous Tolerance Scores: Erythema (assessing skin redness), from Baseline to Day 28. Scale range is 0-3 where 0 = no redness, 1 = mild redness, 2 = moderate redness, and 3 = severe redness.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 43
Units on a scale | -0.07 (0.34)

2. Primary Outcome: Cutaneous Tolerance Scores: Dryness/Scaling
Description: Cutaneous Tolerance Scores: Dryness/Scaling (assessing skin dryness), from Baseline to Day 28. Scale range is 0-3, where 0 = no dryness, 1 = mild dryness, 2 = moderate dryness, and 3 = severe dryness.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 43
Units on a scale | -0.14 (0.41)

3. Primary Outcome: Cutaneous Tolerance Scores: Edema
Description: Cutaneous Tolerance Scores: Edema (assessing skin edema/swelling), from Baseline to Day 28. Scale range is 0-3 where 0 = no edema, 1 = mild edema, 2 = moderate edema, and 3 = severe edema.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 43
Units on a scale | 0.00 (0.00)

4. Primary Outcome: Cutaneous Tolerance Scores: Burning/Stinging
Description: Cutaneous Tolerance Scores: Burning/Stinging (assessing skin burning/stinging), from Baseline to Day 28. Scale range is 0-3 where 0 = no burning/stinging, 1 = mild burning/stinging, 2 = moderate burning/stinging, and 3 = severe burning/stinging.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 43
Units on a scale | 0.00 (0.00)

5. Primary Outcome: Cutaneous Tolerance Scores: Itching
Description: Cutaneous Tolerance Scores: Itching (assessing skin itching), from Baseline to Day 28. Scale range is 0-3 where 0 = no itching, 1 = mild itching, 2 = moderate itching, and 3 = severe itching.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 43
Units on a scale | 0.00 (0.00)

6. Primary Outcome: Cutaneous Tolerance Scores: Tightness/Dry Feeling
Description: Cutaneous Tolerance Scores: Tightness/Dry Feeling (assessing skin tightness/dry feeling), from Baseline to Day 28. Scale range is 0-3 where 0 = no tightness/dry feeling, 1 = mild tightness/dry feeling, 2 = moderate tightness/dry feeling, and 3 = severe tightness/dry feeling.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 43
Units on a scale | -0.05 (0.21)

7. Secondary Outcome: Cutaneous Tolerance Scores: Erythema
Description: Cutaneous Tolerance Scores: Erythema (assessing skin redness), from Baseline to Day 14. Scale range is 0-3 where 0 = no redness, 1 = mild redness, 2 = moderate redness, and 3 = severe redness.
Time Frame: Baseline to Day 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Units on a scale | -0.09 (0.29)

8. Secondary Outcome: Cutaneous Tolerance Scores: Dryness/Scaling
Description: Cutaneous Tolerance Scores: Dryness/Scaling (assessing skin dryness), from Baseline to Day 14. Scale range is 0-3, where 0 = no dryness, 1 = mild dryness, 2 = moderate dryness, and 3 = severe dryness.
Time Frame: Baseline to Day 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Units on a scale | -0.11 (0.44)

9. Secondary Outcome: Cutaneous Tolerance Scores: Edema
Description: Cutaneous Tolerance Scores: Edema (assessing skin edema/swelling), from Baseline to Day 14. Scale range is 0-3 where 0 = no edema, 1 = mild edema, 2 = moderate edema, and 3 = severe edema.
Time Frame: Baseline to Day 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Units on a scale | 0.00 (0.00)

10. Secondary Outcome: Cutaneous Tolerance Scores: Burning/Stinging
Description: Cutaneous Tolerance Scores: Burning/Stinging (assessing skin burning/stinging), from Baseline to Day 14. Scale range is 0-3 where 0 = no burning/stinging, 1 = mild burning/stinging, 2 = moderate burning/stinging, and 3 = severe burning/stinging.
Time Frame: Baseline to Day 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Units on a scale | 0.02 (0.15)

11. Secondary Outcome: Cutaneous Tolerance Scores: Itching
Description: Cutaneous Tolerance Scores: Itching (assessing skin itching), from Baseline to Day 14. Scale range is 0-3 where 0 = no itching, 1 = mild itching, 2 = moderate itching, and 3 = severe itching.
Time Frame: Baseline to Day 14
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Units on a scale | 0.04 (0.21)

12. Secondary Outcome: Cutaneous Tolerance Scores: Tightness/Dry
Description: Cutaneous Tolerance Scores: Tightness/Dry Feeling (assessing skin tightness/dry feeling), from Baseline to Day 14. Scale range is 0-3 where 0 = no tightness/dry feeling, 1 = mild tightness/dry feeling, 2 = moderate tightness/dry feeling, and 3 = severe tightness/dry feeling.
Time Frame: Baseline to Day 14
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Acne Mask
Number analyzed (Participants) | 45
Units on a scale | -0.02 (0.26)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time a signed and dated informed consent was obtained at Baseline until Day 28 or subject's last visit. Serious adverse events were also reportable within 30 calendar days of subject's last visit. Spontaneously reported seriously adverse events after the 30 calendar days period assessed by the investigator to be study related would be reportable to the Sponsor.
Description: The investigator or a designee interviewed subjects for changes in health/medication at each visit, documenting any reported adverse events.
Arm/Group | Acne Mask
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for any public disclosure of the data or results, the PI will provide the Sponsor with at least 60 days for review of the publication. Sponsor's written consent is required for any publication containing the Sponsor's confidential information. The Sponsor may request that the PI withholds such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03128723/Prot_SAP_000.pdf